CLINICAL TRIAL: NCT00909714
Title: Neuroregeneration Enhanced by TDCS in Stroke
Brief Title: Neuroregeneration Enhanced by Transcranial Direct Current Stimulation (TDCS) in Stroke
Acronym: NETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NETS Trial
Record Dates: First submitted 2009-05-12; First posted 2009-05-28 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: stroke; non-invasive cortical stimulation; motor recovery; cortical plasticity; TDCS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anodal tDCS (Experimental): Direct Current (DC)-Stimulator to apply tDCS + Training
  Interventions: Device: DC-Stimulator to apply tDCS
- Sham tDCS (Sham Comparator): Direct Current (DC)-Stimulator to apply Sham tDCS (Placebo) + Training
  Interventions: Device: DC-Stimulator to apply Sham tDCS

INTERVENTIONS:
Device: DC-Stimulator to apply tDCS — Anodal tDCS (20 minutes) stimulation will be applied once a day in combination with standardized upper extremity rehabilitative training
  Arms: Anodal tDCS
Device: DC-Stimulator to apply Sham tDCS — Sham stimulation will be applied once a day in combination with standardized upper extremity rehabilitative training
  Arms: Sham tDCS

SUMMARY:
Testing the hypothesis that non-invasive brain stimulation by transcranial direct current stimulation (tDCS) combined with functional training in the subacute phase of first-ever stroke will enhance functional regeneration compared with a Placebo intervention.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability, which significantly impairs the economic and social life of patients and society. Every year 200 000 to 250 000 patients suffer a stroke in Germany. Only a small number of the stroke survivors recover to a degree that allows them to return into their professional and private life. Despite significant efforts to develop novel and efficient treatment strategies the level of functional regeneration is still not satisfying. Thus, the development of innovative and effective treatment strategies will have a major impact for the patients' life, the society and the public health system.

Within the proposed project an innovative, non-invasive and cost effective interventional strategy, based on the combination of a specific rehabilitative training and brain stimulation by transcranial direct current stimulation (tDCS), will be used to enhance functional regeneration in stroke patients. The intervention will be applied in an early stage in which plasticity, cortical reorganization and functional improvement is most pronounced. We hypothesize that the combination of anodal tDCS delivered to the motor cortex of the affected hemisphere combined with training over a period of two weeks in the subacute stage after stroke will significantly enhance cortical plasticity, functional regeneration and long-term outcome determined by clinical and functional outcome measures compared with Placebo stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subacute stroke patients (5-45 days after stroke) with thromboembolic non-hemorrhagic subcortical or cortical, first clinically overt stroke will be included. Moderate to moderately severe upper-extremity hemiparesis, defined as an Upper Extremity Fugl-Meyer score (UEFMA) between 20 and 58 (inclusive).

Exclusion Criteria:

* pre-existing large lesions (> 1.5 cm maximum diameter) in a brain area that belongs to the anatomically established sensorimotor/premotor system
* progressive stroke
* completely lesioned hand knob area of M1 affected if no motor evoked potentials (MEPs) elicited by transcranial magnetic stimulation (TMS) are present
* bilateral motor impairment
* florid alcohol and/or drug abuse
* florid severe psychiatric illness (e.g. schizophrenia)
* severe language disturbances that prevents the patient to give informed consent or inhibit adequate scoring because of insufficient understanding of scoring introductions
* tumor diseases with a life expectancy less than one year
* increased intracranial pressure
* polyneuropathy and/or ischemic peripheral disease if the sensorimotor functions of the upper extremities are affected clinically relevant
* severe cognitive deficits (MMSE ≤ 23)
* pregnancy
* contraindication for MRI or TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer-Assessment (UEFMA) | 1-7 days after the end of the intervention
  standardized test of upper extremity function

SECONDARY OUTCOMES:
Upper Extremity Fugl-Meyer-Assessment (UEFMA) | 30±10 days after the intervention
  standardized test of upper extremity function
Upper Extremity Fugl-Meyer-Assessment (UEFMA) | 90±20 days after the intervention
  standardized test of upper extremity function
Upper Extremity Fugl-Meyer-Assessment (UEFMA) | Long-term outcome | 12±1 months after the intervention
  standardized test of upper extremity function
Action Research Arm Test (ARAT) | 1-7 days after the end of the intervention
  standardized tests of upper extremity function
Action Research Arm Test (ARAT) | 30±10 days after the intervention
  standardized tests of upper extremity function
Action Research Arm Test (ARAT) | 90±20 days after the intervention
  standardized tests of upper extremity function
Action Research Arm Test (ARAT) | Long-term outcome | 12±1 months after the intervention
  standardized tests of upper extremity function
Nine Hole Peg Test (NHPT) | 1-7 days after the end of the intervention
  standardized test to assess fine motor skills
Nine Hole Peg Test (NHPT) | 30±10 days after the intervention
  standardized test to assess fine motor skills
Nine Hole Peg Test (NHPT) | 90±20 days after the intervention
  standardized test to assess fine motor skills
Nine Hole Peg Test (NHPT) | Long-term outcome | 12±1 months after the intervention
  standardized test to assess fine motor skills
Stroke Impact Scale (SIS) | 1-7 days after the end of the intervention
  questionnaire is to evaluate how stroke has impacted health and life of patients
Stroke Impact Scale (SIS) | 30±10 days after the intervention
  questionnaire is to evaluate how stroke has impacted health and life of patients
Stroke Impact Scale (SIS) | 90±20 days after the intervention
  questionnaire is to evaluate how stroke has impacted health and life of patients
Stroke Impact Scale (SIS) | Long-term outcome | 12±1 months after the intervention
  questionnaire is to evaluate how stroke has impacted health and life of patients
Box-and-Block Test | 1-7 days after the end of the intervention
  standardized test to assess fine motor skills
Box-and-Block Test | 30±10 days after the intervention
  standardized test to assess fine motor skills
Box-and-Block Test | 90±20 days after the intervention
  standardized test to assess fine motor skills
Box-and-Block Test | 12±1 months after the intervention
  standardized test to assess fine motor skills
Grip Force | 1-7 days after the end of the intervention
  dynamometer-based test to assess grip strength
Grip Force | 30±10 days after the intervention
  dynamometer-based test to assess grip strength
Grip Force | 90±20 days after the intervention
  dynamometer-based test to assess grip strength
Grip Force | 12±1 months after the intervention
  dynamometer-based test to assess grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gerloff, Prof. Dr., Principal Investigator — Department of Neurology, University Medical Center Hamburg-Eppendorf
Locations (11):
- Neurologische Universitätsklinik Wien, Vienna, Vienna, Austria
- Germany (9):
  - Klinik Kipfenberg, Kipfenberg, Bavaria
  - Brandenburgklinik Berlin-Brandenburg, Bernau Bei Berlin, State of Berlin
  - Neurologie Moritzklinik, Bad Klosterlausnitz, Thuringia
  - Neurologische Klinik Bad Aibling, Bad Aibling
  - Neurologisches Zentrum Segeberger Kliniken, Bad Segeberg
  - NRZ Leipzig, Bennewitz
  - MEDIAN Klinik Berlin-Kladow, Berlin
  - University Medical Center Hamburg Eppendorf (UKE), Hamburg
  - University Medical Center Heidelberg, Heidelberg
- Fondazione Santa Lucia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is planned after main publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: Within 24 months after main publication.
Access Criteria: Personal login into UKE data repository.

REFERENCES:
- [Background] NETS Trial Collaboration Group. A multicenter, randomized, double-blind, placebo-controlled trial to test efficacy and safety of transcranial direct current stimulation to the motor cortex after stroke (NETS): study protocol. Neurol Res Pract. 2022 Apr 18;4(1):14. doi: 10.1186/s42466-022-00171-2. PMID 35430801
- [Background] NETS Trial Collaboration Group. Efficacy and safety of transcranial direct current stimulation to the ipsilesional motor cortex in subacute stroke (NETS): a multicenter, randomized, double-blind, placebo-controlled trial. Lancet Reg Health Eur. 2024 Jan 2;38:100825. doi: 10.1016/j.lanepe.2023.100825. eCollection 2024 Mar. PMID 38476746
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411